CLINICAL TRIAL: NCT04303533
Title: Regulation of Amygdala Via Neurofeedback in PTSD After Childhood Sexual Abuse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0576-18
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: PTSD
Keywords: Neuro-Feedback; Childhood Sexual Abuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EFP-NF (Experimental)
  Interventions: Device: Neuro-Feedback EFP

INTERVENTIONS:
Device: Neuro-Feedback EFP — Neurofeedback (NF) - is a treatment method based on learned self-modulation of neural activity in response to feedback of neural signal. Amygdala-EFP (EEG-finger-print, EFP) is an EEG-NF application that modulates amygdala response.

SUMMARY:
Post-traumatic stress disorder (PTSD) is a common debilitating disorder that affects many individuals exposed to aversive events. The severity of PTSD symptoms is positively correlated with amygdala activation. More severe PTSD symptoms following exposure to stressful events, are associated with amygdala hyper-responsivity prior to exposure. A possible intervention for PTSD is Neurofeedback (NF) - a treatment method based on learned self-modulation of neural activity in response to feedback of neural signal. Previous work in the investigator's lab established a NF training procedure that utilizes the temporal abilities of EEG with the spatial advantages of fMRI. Further work based on this method using the amygdala BOLD signal (EEG-finger-print, EFP) has demonstrated a potential for improving the ability to self-regulate amygdala activity and to improve emotional regulation in a healthy population. The current study aims to investigate the potential of this method as a therapeutic intervention for PTSD among men with a history of childhood sexual abuse (CSA).

DETAILED DESCRIPTION:
Pretreatment phase- All participants will undergo clinician evaluation and self-report measures in TASMC. In addition, they will receive a WatchPAT (wearable technology) for tracking sleep for 2 nights.

Participants will receive 10 sessions of NF-EFP once a week for ten weeks. NF-EFP sessions: For the duration of each NF-EFP session the participant will be seated comfortably in front of a computer screen. A staff member will explain the goal of the meeting to the participant, present the equipment to be used and describe the course of the meeting. The EEG-NF practice will consist of four-minute segments repeated for up to 30 minutes. During each practice segment the participant will be asked to modify visual media that provides feedback on the degree of successful brain training. The duration of one session is approximately 45 minutes.

Post treatment phase -All participants will undergo clinician evaluation and self-report measures in TASMC. In addition, they will receive a WatchPAT (wearable technology) for tracking sleep for 2 nights.

ELIGIBILITY:
Inclusion Criteria:

Treated at Clinic for Sexual Assault with stable symptoms. Fulfill screening criteria of DSM-V for PTSD.

-

Exclusion Criteria:

* Fulfill screening criteria of DSM-V for psychosis. Substance dependence or abuse other than nicotine. Diagnosis of a neurodegenerative disease. Acute illness that could be worsen by the treatment. -

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 4 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical measures- PSTD symptoms | [ Time Frame: The clinical assessment will be administrated at pre-treatment (baseline) and post-treatment (up to two weeks post-treatment)
  Change in PTSD symptoms measured by change in Clinician-Administered PTSD Scale (CAPS)

SECONDARY OUTCOMES:
Sleep quality- REM latency and sleep latency | [ Time Frame: Two nights; first, at pre-treatment (baseline) and second, post-treatment (up to two weeks post-treatment).
  WatchPAT (wearable technology) will track REM latency and sleep latency . These will be compared and corrected using MANOVA as an outcome analysis. To assess sleep globally, we will aggregated: increased sleep latency , reduced sleep efficiency (the ratio of the total time spent asleep compared to the total amount of time spent in bed) and lack of proper deep sleep (quantified using "deep sleep percent" and "REM sleep percent", i.e. the ratio of the total time spent in deep/REM sleep out of the total sleep time) into one reported value. For full explanation and calculation of index see Goldway, et al. (2019).
Self-report questionnaires- PCL (PTSD checklist ) | The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).
  A self-report measure (20 items) of PTSD symptoms reflecting the diagnostic criteria of DSM 4+5. The self-report rating scale is 0-4 for each symptom, Rating scale descriptors are: "Not at all," "A little bit," Moderately," "Quite a bit," and "Extremely." A total symptom severity score (range - 0-80) is obtained by summing the scores for each of the items, higher values represent more severe PTSD. Symptom cluster severity scores is obtained by summing the scores for the items within a given cluster, i.e. for DSM 5: cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20).
self-report questionnaires- Beck Depression Inventory (BDI-II) | Time Frame: The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).
  A 21 item self-administered inventory of depression symptoms and their respective intensity. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The maximum total score is 63. higher values represent more severe depression.
Self-report questionnaires- State-trait Anxiety Inventory (STAI) | Time Frame: The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).
  A 20 item self-administered inventory of state and trait anxiety. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). SUM of scores is obtained, higher scores indicate greater anxiety.
Self-report questionnaires- Toronto Alexithymia Scale (TAS) | Time Frame: The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment)
  20 items self-administered composing the alexithymia scale. The TAS-20 has 3 sub-scales: Difficulty Describing Feelings subscale is used to measure difficulty describing emotions. Difficulty Identifying Feeling subscale is used to measure difficulty identifying emotions. Externally-Oriented Thinking subscale is used to measure the tendency of individuals to focus their attention externally. Items are rated using a 5-point Likert scale whereby 1 = strongly disagree and 5 = strongly agree. The total alexithymia score is the sum of responses to all 20 items, while the score for each subscale factor is the sum of the responses to that subscale. Higher scores represent higher alexithymia rate.
Self-report questionnaires- Dissociative Experience Scale (DES) | ime Frame: The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).
  28-item self-administered measure of frequency of dissociative experiences. higher DES scores indicate higher dissociative rates.
Self-report questionnaires- Locus of Control (LOC) | ime Frame: The Self-report questionnaires will be administrated: pre-treatment (baseline), post-treatment (up to two weeks post-treatment).
  24 items self-administered questionnaire intended to measure internal versus external locus of control

IPD SHARING:
Plan to Share IPD: No